CLINICAL TRIAL: NCT06298136
Title: The Effects of an Online Mindfulness-based Intervention for Parents of Children with Attention-Deficit/Hyperactivity Disorder: a Randomized Controlled Trial
Brief Title: The Effects of an Online Mindfulness-based Intervention for Children with Attention-Deficit/Hyperactivity Disorder
Acronym: MindADHD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, LO Hay-ming Herman, Associate Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15610923
Record Dates: First submitted 2024-02-22; First posted 2024-03-07 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-02

CONDITIONS: ADHD
Keywords: ADHD; family; mindfulness-based intervention; online intervention; randomized controlled trial
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: This study will investigate the effects of an online mindfulness-based intervention (MBI) on outcomes in children with ADHD. The effects of the MBI (arm 1) will be investigated in comparison with the effects of psychoeducation (arm 2).
Who Masked: Participant, Outcomes Assessor
Masking Description: The participants will be informed that an intervention (program A or program B) will be assigned to them randomly. For research team who will be in contact with participants for outcome assessment, whether the participants have been allocated to arm 1 or arm 2 will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Online mindfulness-based intervention (MBI) (Experimental): The research team have developed an online family MBI (arm 1) for parents and their children with ADHD. It integrates psychoeducation videos (each 3-7 minutes) with audio mindfulness exercises (each 5-15 minutes). The content includes: (1) mindfulness and attention, (2) mindfulness and physical sensation, (3) mindfulness and parental stress, and (4) mindfulness and parental self-care. The majority of the exercises in the first four modules are for parents, but five of them include guidance for child-parent mindfulness exercises. The fifth module targets children with ADHD and the length of video and audio of mindfulness exercises for children, each last 3-5 mins.
  Interventions: Behavioral: mindfulness-based intervention
- Psychoeducation (Active Comparator): The psychoeducation program is based on the Parent Training for Child ADHD Program developed by Russell Barkley for children with ADHD and other behavioral disorders. It includes: (1) understanding ADHD symptoms, (2) general behavior management principles, (3) positive reinforcement and attending skills, (4) the use of a reward and token system, and (5) child problem-solving skills.
  Interventions: Behavioral: child behavior management

INTERVENTIONS:
Behavioral: mindfulness-based intervention — Audio exercises as homework assignment will be included. Four instructor-led online real time sessions are provided
  Arms: Online mindfulness-based intervention (MBI)
Behavioral: child behavior management — worksheet will be provided to guide parents and children in behavior change. Four instructor-led online real time sessions are provided.
  Arms: Psychoeducation

SUMMARY:
This study will investigate the effects of an online mindfulness-based intervention with a randomized controlled trial.

DETAILED DESCRIPTION:
In Hong Kong, 3.9% of adolescents were diagnosed as having Attention Deficit/Hyperactivity Disorder (ADHD). The primary symptoms of ADHD include inattention, hyperactivity, and impulsivity, which limit learning and socioemotional development. ADHD has been associated with poor family functioning, increased stress within the family, higher rates of parental psychopathology, and conflicted parent-child relationships. More than 70% of children with ADHD experience improvements after treatment with psychostimulant medication but some children demonstrate side effects. Behavioral interventions have been found to be effective in enhancing motivation and decreasing the disruptive behaviors of children with ADHD. However, some parents of children with ADHD experience high levels of stress, and the children's symptoms and reactions often complicate their application of the techniques taught in parent behavioral training programs. Moreover, while children benefit from behavioral training in short-term improvements, its long-term effects are uncertain, as children with ADHD cannot learn self-regulation without parental supervision.

In recent reviews and randomized controlled trials, mindfulness-based intervention (MBI) has shown its benefits in improving ADHD symptoms and parent's mental health. Practitioners and researchers have collaborated to apply technology and convert face-to-face MBIs into online or app-based MBIs. Our research team modified the ordinary MBI program structure by integrating short daily online psychoeducation videos with audio mindfulness guidance. In view of the poor engagement and high dropout issues of many online programs, our program is strengthened by incorporating four weekly, real-time online meetings with instructors. The content of MBI includes mindfulness and attention, mindfulness and physical sensation, mindfulness and parental stress, and mindfulness and self-care. The majority of the exercises are for parents, but additional guidance for child-parent mindfulness exercises is included. One module will target children with ADHD and the length of video and audio of mindfulness exercises for children.

This study will investigate the effects of an online MBI, with a randomized controlled trial. A total of 208 parents will be recruited, and randomly assigned to online MBI and psychoeducation. The effects of the MBI will be investigated in comparison with the effects of psychoeducation and outcomes on child ADHD symptoms, parent mental health, and family expressed emotions will be measured. Immediate effect at post-intervention, and 3-month follow-up maintenance effect will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* parents of children diagnosed with ADHD by a psychiatrist and psychologist according to the Diagnostic and Statistical Manual of Mental Disorders, 5th Ed (DSM-5)
* parents of children with ADHD aged 6 to 12.
* Parents who have served as the primary caregivers of their children in the last year and children with ADHD who speak and understand Cantonese Chinese.
* Children either not taking any medication or maintaining a stable dosage of the same ADHD medication for at least 3 months prior to study enrollment and having no plans to change medication and dosage during the study period.

Exclusion Criteria:

* parents diagnosed with developmental disabilities, psychosis, or cognitive impairment, who may thus have difficulty comprehending the content of the project.
* Children with another developmental disability such as autistic spectrum disorder or intellectual disability.
* Parents who completed an eight-week MBI or equivalent program.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 208 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Child ADHD symptoms | Change from pre-intervention, to 1-month follow-up, and 3-month follow-up
  Strengths and Weaknesses of ADHD Symptoms and Normal Behaviors rating Scale, minimum value is -54 and maximum value is 54. The higher the score, the severe the symptoms of inattention and hyperactivity.

SECONDARY OUTCOMES:
Parent depressive symptoms | Change from pre-intervention, to 1-month follow-up, and 3-month follow-up
  The Center for Epidemiologic Studies Depression Scale. minimum value is 0 and the maximum value is 30. The higher the score, the severe the symptoms of depression.
Parent anxiety symptoms | Change from pre-intervention, to 1-month follow-up, and 3-month follow-up
  Hospital Anxiety and Depression Scale - Anxiety subscale. minimum value is 0 and the maximum value is 21. The higher the score, the severe the symptoms of anxiety.
Parent sleep quality | Change from pre-intervention, to 1-month follow-up, and 3-month follow-up
  Insomnia Severity Index. minimum value is 0 and the maximum value is 28. The higher the score, the severe the symptoms of sleep quality.
Parent well-being | Change from pre-intervention, to 1-month follow-up, and 3-month follow-up
  World Health Organization Well-Being Index. minimum value is 0 and the maximum value is 25. The lower the score, the worse in well-being.
Child executive functioning | Change from pre-intervention, to 1-month follow-up, and 3-month follow-up
  Behavior Rating Inventory of Executive Function (second edition). minimum value is 0 and the maximum value is 126. The higher the score, the severe the deficits in executive functioning.
Parental Stress | Change from pre-intervention, to 1-month follow-up, and 3-month follow-up
  Parenting Stress Index (short form). minimum value is 36 and the maximum value is 180. The higher the score, the severe the parenting stress.
Expressed emotion | Change from pre-intervention, to 1-month follow-up, and 3-month follow-up
  The Five Minute Speech Sample. It is scored by the coding procedure. There is no maximum value. THe higher the score, the severe the parent's expressed emotion.

CONTACTS AND LOCATIONS:
Overall Officials: Herman Hay Ming Lo, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- Herman Hay Ming Lo, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
The study protocol will be published. The data collected in this study excluding personal data can be shared by sending request to principal investigator.
Supporting Information: Study Protocol, SAP
Time Frame: The protocol will be submitted for publication within 2024. The data collected in this study will be shared after the publication of the study is published.
Access Criteria: Individuals who request the data should indicate the purpose clearly when submitting their requests.